CLINICAL TRIAL: NCT00229463
Title: Study of Genetic Differences in People With Depression
Acronym: Genetics
Status: Completed | Type: Observational
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Andrew F. Leuchter, Principal Investigator, University of California, Los Angeles
Other Study IDs: 01-10-049
Record Dates: First submitted 2005-09-28; First posted 2005-09-29 (Estimated); Last update posted 2016-11-18 (Estimated); Status verified 2016-10

CONDITIONS: Depressive Disorder, Major
Keywords: Depression; genetic; gene; antidepressant; research
MeSH Terms: conditions — Depressive Disorder, Major; Depression

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to identify genes involved in depression. Specifically, the investigators will analyze some genes that may be related to whether or not a person responds to antidepressant medication. This project is part of basic scientific research to increase understanding of the role of genetic influences in psychological and mental processes involved in the response to treatment for depression.

ELIGIBILITY:
Inclusion Criteria:

* History of Unipolar Major Depression
* Control subjects must be healthy normal adults

Exclusion Criteria:

* Subjects with mood symptoms that are not severe enough to qualify for MDD
* Subjects with any active medical illness that may be related to ongoing mood disorder
* Normal subjects must be free from: a psychiatric diagnosis, substance abuse, a history of seizure disorder, and any serious medical illness

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited from previous studies conducted at the Laboratory of Brain, Behavior, and Pharmacology, where subjects' response to treatment has already been determined. This strategy offers the advantage that no new subjects need to be enrolled in placebo-controlled treatment studies.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2002-01; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew F. Leuchter, M.D., Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA Semel Institute for Neuroscience and Human Behavior, Los Angeles, California, United States

REFERENCES:
- See also: Depression Research - Click here for more information about this study: Study of Genetic Differences in People with Depression — http://www.DepressionResearch.com/